CLINICAL TRIAL: NCT00709254
Title: Phase I, 3-Period, Fasting, Bioavailability, Safety Assessment and PK Study Evaluating Single Dose Administration of i.v. Fentanyl (200 µg) and Single and Multiple Doses of 3 mL of Inhaled AeroLEF (Liposome-Encapsulated Fentanyl 500 µg/mL) Administered in Normal Healthy Subjects
Brief Title: Study of Single and Multiple Doses of Inhaled AeroLEF (Liposome-Encapsulated Fentanyl)in Healthy Subjects
Acronym: LEF-2495
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Responsible Party: Ali Raza, Chief Medical Officer, YM BioSciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LEF-2495
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
Keywords: AeroLEF; fentanyl; pharmacokinetics; liposome; encapsulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group A (Active Comparator): Subjects received an i.v. dose of fentanyl (200 µg)
  Interventions: Drug: i.v. fentanyl
- Treatment Group B (Experimental): Subjects received a single dose of 3 mL AeroLEF (500 µg/1 mL)
  Interventions: Drug: 3 mL AeroLEF (500 µg/1 mL)
- Treatment Group C (Experimental): Subjects received multiple doses of 3 mL AeroLEF (500 µg/1 mL) every 12 hours for a total of five doses over a 3 days
  Interventions: Drug: 3 mL AeroLEF (500 µg/1 mL)

INTERVENTIONS:
Drug: i.v. fentanyl — single dose, 200 ug
  Other Names: fetanyl citrate injection
  Arms: Treatment Group A
Drug: 3 mL AeroLEF (500 µg/1 mL) — A single dose of 3mL (500 µg/1 mL) of AeroLEF (Aerosolized Free and Liposome-Encapsulated Fentanyl)
  Other Names: Aerosolized Free and Liposome-Encapsulated Fentanyl
  Arms: Treatment Group B
Drug: 3 mL AeroLEF (500 µg/1 mL) — A multiple doses of 3mL (500 µg/1 mL)of AeroLEF (Aerosolized Free and Liposome-Encapsulated Fentanyl)every 12 hours for a total of five doses over a 3 days
  Other Names: Aerosolized Free and Liposome-Encapsulated Fentanyl
  Arms: Treatment Group C

SUMMARY:
This study was designed to assess single-dose and multiple-dose PK and safety parameters utilizing a dosage of 3 mL (500 µg/mL)AeroLEF delivered via nebulization with the AeroEclipse BAN device. The study was conducted in opioid naïve subjects who were not blocked with naloxone or other opioid receptor antagonists.

DETAILED DESCRIPTION:
Period I: Subjects received an i.v.dose of fentanyl (200 µg) (Treatment A).

Period II: Subjects were randomly assigned to receive either a single-dose (Treatment B) or multi-dose (Treatment C) of AeroLEF.

In the multi-dose Treatment C group, subjects received a dose of 3 mL AeroLEF every 12 hours for a total of five doses over a 3 days with a 4 week washout period before crossing over to Period III.

Period III: Subjects from Period II participated in the crossover study and receive either a multi-dose (Treatment C, 5 doses at 12 hour intervals) or a single dose (Treatment B). Subjects in Treatment B or Treatment C were instructed to continue inhalation of AeroLEF for approximately one (1) minute beyond the point of nebulizer sputter to ensure that all aerosolized medication was delivered.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female with a minimum age of at least 18 years
* Body weight with aBMI range of 18.5 - 27, with a minimum weight of at least 60 kg.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed, written, Informed Consent Form.
* Normal findings in the physical examination, vital signs (blood pressure between 100-140 - 60-90 mmHg, heart rate between 55-99 beats/min, respiration rate between 12-20 minute) and a 12 lead ECG.
* Negative for drug abuse, nicotine, alcohol, hepatitis B-surface antigen, hepatitis C and HIV.
* If a female of child-bearing potential, the patient must have a negative urine pregnancy test at screening and baseline.
* No clinical laboratory values outside of the Principal Investigator's acceptable range, unless the Principal Investigator decided that the subject's values are not clinically significant.
* Female subjects: (a) if pre-menopausal, have regular menstrual cycles (28-32 days), and (b) are not pregnant prior to study start and avoids pregnancy during the study and 1 month post drug administration, or (c) were surgically sterile for at least 6 months prior to enrollment, or (d) are post-menopausal for at least 1 year prior to enrollment.

Exclusion Criteria:

* Known history of hypersensitivity to fentanyl.
* Presence or history of cardiac, pulmonary, gastrointestinal, endocrine, neuromuscular, neurologic, hematological, liver or kidney disease, or any condition known to interfere with absorption, distribution , metabolism, or excretion of drugs.
* History of drug abuse or narcotic dependency.
* Use of prescription medication within 30 days preceding entry int the study, including any enzyme inducing/inhibitory drugs (excluding contraceptives).
* Participating in a clinical trial with an investigational drug within 30 days preceding this trial.
* Blood donation within 45 days preceding this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-12; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | continuously

SECONDARY OUTCOMES:
pharmacokinetics and bioavailability | various time points

CONTACTS AND LOCATIONS:
Overall Officials: Diana Pilura, PhD, Study Director — YM BioSciences; Paul Y Tam, MD, FACP, Principal Investigator — University of Toronto, Ontario, Canada
Locations (1):
- University of Toronto, Toronto, Ontario, Canada